CLINICAL TRIAL: NCT06141421
Title: A Real-World Study to Evaluate the Clinical Performance and Safety of da Vinci SP Surgical System for Single-Port Colorectal Surgeries
Brief Title: A Real-World Study to Evaluate the Clinical Performance and Safety of da Vinci SP Surgical System for Single-Port Colorectal Surgeries（SPiM-RWS-CR）
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Ren, Pro.Zhao, Ruijin Hospital
Other Study IDs: ISFMT-SP-003
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Single-Port Colorectal Surgeries
Keywords: Single-Port Colorectal Surgeries; low anterior resection of the rectum with or without total mesorectal excision; right hemicolectomy, left hemicolectomy and sigmoidectomy with or without transanal total mesocolic excision and central blood vessel ligation; transanal minimally invasive surgery
MeSH Terms: interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- RWS study for SP CR Surgeries da Vinci SP Surgical System(SP1098)
  Interventions: Procedure: procedure

INTERVENTIONS:
Procedure: procedure — procedure

SUMMARY:
A real-world study to evaluate the clinical performance and safety of da Vinci SP Surgical System ("SP single-port robot" for short) for single-port robot-assisted colorectal surgeries in the real world, providing a real world evidence for clinical application of the product in the Chinese population.

English name: da Vinci SP Surgical System Model and specification: SP1098 Manufacturer: Intuitive Surgical, Inc.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have received or plan to receive colorectal surgeries with the SP single-port robot, such as low anterior resection of the rectum with or without total mesorectal excision; right hemicolectomy, left hemicolectomy and sigmoidectomy with or without transanal total mesocolic excision and central blood vessel ligation; and transanal minimally invasive surgery.
2. Patients who voluntarily decide to participate in the study and sign the ICF (or exempt from signature of the ICF as approved by the EC).

Exclusion Criteria:

1. Patients with missing data on the primary endpoint in retrospective cases;
2. Subjects having any contraindications of single-port robot surgery;
3. The intraoperative anatomy determined that minimally invasive surgery was not suitable;
4. Patients who are considered inappropriate to participate in this study by investigator.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have received or plan to receive colorectal surgeries with the SP single-port robot, such as low anterior resection of the rectum with or without total mesorectal excision; right hemicolectomy, left hemicolectomy and sigmoidectomy with or without transanal total mesocolic excision and central blood vessel ligation; and transanal minimally invasive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Intraoperative conversion rate | Intraoperative
The incidence of device-related or likely related complications of Clavien-Dindo classification grade III or higher at postoperative 30 days | 30 days

SECONDARY OUTCOMES:
Intraoperative bleeding volume | Intraoperative
The rate of intraoperative blood transfusion | Intraoperative
Surgical duration | Intraoperative
Length of stay (LOS) | During the follow-up 1 day before discharge
Admission to ICU and ICU LOS | During the follow-up 1 day before discharge
Urethral catheter indwelling duration | in the follow-up 1 month after the surgery
Postoperative pain score | follow-ups 1 day (24±4 h), 3 days (72±4 h) and 1 month (30±5 days) after the surgery.
Short-term recovery of functions | in the follow-up 1 month after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided